CLINICAL TRIAL: NCT03354832
Title: Research Action on Infant Mortality in Reunion Island Evaluation of Factors Affecting In-utero Foetal Death and New-born Death in Reunion Island
Brief Title: In-utero Death and Birth Mortality in Reunion Island
Acronym: RAMIR
Status: Terminated | Type: Observational
Why Stopped: small number of utero death, mothers refused to participate
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/CHU/08
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Pregnancy Loss; Infant Death
MeSH Terms: conditions — Infant Death | interventions — Contraception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Foetal death: In-utero dead foetus weighting at least 500 g or 22-amenorrhea weeks old. In utero death means that death occurs during delivery or per partum
  Interventions: Other: Foetal death
- New-born death: New-born dead during post-birth hospital stay and at least 23-amenorrhea weeks old.
  Interventions: Other: New-born death
- Birth control for foetal death: Same gender child born, and alive, in the same hospital, and born on time (37-41 amenorrhea weeks old).
  Interventions: Other: Birth control for foetal death
- Birth control for new-born death: Same gender infant born, and alive, in the same hospital, and:
  * for 23-amenorrhea weeks old new-born death: control new-born are born on time (37-41 amenorrhea weeks old).
  * for 24 to 31-amenorrhea weeks old new-born death: control new-born are premature infant (24-31 amenorrhea weeks old), and are included when their hospital stay ends.
  * for 32 and more-amenorrhea weeks old new-born death: control new-born are 32 and more-amenorrhea weeks old infant
  Interventions: Other: Birth control for new-born death

INTERVENTIONS:
Other: Foetal death — A midwife is in charge to interview the mother during the month following the lost of her infant.
  Groups: Foetal death
Other: New-born death — A midwife is in charge to interview the mother during the month following the lost of her infant.
  Groups: New-born death
Other: Birth control for foetal death — A midwife is in charge to interview the mother during her hospital stay
  Groups: Birth control for foetal death
Other: Birth control for new-born death — A midwife is in charge to interview the mother during her hospital stay
  Groups: Birth control for new-born death

SUMMARY:
Infant mortality is still relevant despite the improvement and the accessibility of hospital care. Premature birth are two fold higher than in metropolitan France. Some factors has been suspected such as precariousness, alcoholism, congenital malformation, care accessibility, epidemic environment ... Nevertheless, the impact of these factors on foetal death or new-born death are not yet sufficiently quantified to provide appropriate care and prevention action in Reunion Island.

DETAILED DESCRIPTION:
Through the analysis of interview of the mothers that have lost their infant during pregnancy or just after birth, the study aims to draw a picture of the pregnancy cares offer and pregnancy conditions in Reunion Island.

This study is an non interventional case-control study. Socio-economic conditions, pregnancy care and prevention are screened to identified the major cause of foetal or new-born death in Reunion Island. These data are still lacking and will be useful to identify which public health actions that should be organized.

ELIGIBILITY:
Inclusion Criteria:

* Case: foetal death (foetus weighing more than 500 g or more than 22-amenorrhea weeks old) or new-born death (premature: more than 23-amenorrhea weeks old or mature)
* Control: premature (more than 23-amenorrhea weeks old) or mature new-born, alive when the leave the hospital

Exclusion Criteria:

* medical abortion
* second pregnancy during the study period
* case under forensic expertise

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregant women or mother leaving in Reunion Island. Case and control women should have stay during all their pregancy and should have been admitted in an hospital in Reunion Island for delivery.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of suboptimal care | within 4 weeks after birth (control) or lost (case)
  The main suboptimal care are searched:
  * lack or inefficient corticotherapy during pregnancy
  * infant birth in an under equipped hospital, without facilities for premature birth
  * prenatal diagnosis of serious congenital malformations involving specific care at birth
  * lack of B-streptococcus detection
  * unexpected caesarean section during delivery
  * unexpected dystocia

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard GOUYON, Pr, Principal Investigator — Centre Hpospitalier Universitaire de La REUNION
Locations (1):
- Chu Reunion Island, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No